CLINICAL TRIAL: NCT03379389
Title: Clinical Assessment of Urinary Antiseptics Methenamine and Methylthioninium in Recurrent Cystitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundação Educacional Serra dos Órgãos (Other)
Responsible Party: Principal Investigator, Carlos Pereira Nunes, Professor of Internal Medicine, Fundação Educacional Serra dos Órgãos
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AUCR-01-05-17
Record Dates: First submitted 2017-12-08; First posted 2017-12-20 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-11

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections | interventions — Methenamine; Methylene Blue; Acriflavine; Anti-Bacterial Agents; Anti-Infective Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methenamine + Methylthioninium (Experimental): Dosage: Methenamine (120mg) + Methylthioninium (20mg) Dosage form: coated tablets Frequency: 2 coated tablets twice daily Duration: 6 days
  Interventions: Drug: Methenamine + Methylthioninium; Drug: Antibiotics
- Methenamine+Methylthioninium+Acriflavine+Atropa belladona (Active Comparator): Dosage: Methenamine (250mg) + Methylthioninium (20mg) + Acriflavine hydrochloride (15mg) + Atropa belladonna L. (15mg) Dosage form: coated tablets Frequency: 2 coated tablets twice daily Duration: 6 days
  Interventions: Drug: Methenamine + Methylthioninium + Acriflavine + Atropa belladona; Drug: Antibiotics

INTERVENTIONS:
Drug: Methenamine + Methylthioninium — Methenamine + Methylthioninium
  Other Names: methenamine + methylene blue
  Arms: Methenamine + Methylthioninium
Drug: Methenamine + Methylthioninium + Acriflavine + Atropa belladona — Methenamine + Methylthioninium + Acriflavine + Atropa belladona
  Other Names: methenamine + methylene blue + acriflavine + A. belladona
  Arms: Methenamine+Methylthioninium+Acriflavine+Atropa belladona
Drug: Antibiotics — Antibiotics based on individual subjects urine culture / antibiogram
  Other Names: Antimicrobials

SUMMARY:
This is a double-blind, randomized, double-dummy, comparative study in parallel groups of subjects presenting with recurrent cystitis (≥2 episodes within the past 6 months). Subjects will be randomized and treated with one of two presentations of urinary antiseptics containing methenamine and methylthioninium for three days, followed by three days of antibiotic therapy as determined by urine culture and antibiogram. This study aims to assess the efficacy and safety of each treatment.

DETAILED DESCRIPTION:
This is a double-blind, randomized, double-dummy, comparative study in parallel groups of subjects presenting with recurrent cystitis (≥2 episodes within the past 6 months). After initial evaluations including urine culture and antibiogram, a total of 284 subjects will be randomized and treated with one of two presentations of urinary antiseptics containing methenamine and methylthioninium for six days. After three days of treatment, subjects will return to the study center and antibiotic therapy based on the results of the urine culture and antibiogram will be initiated for each subject, to be continued for the remaining three days of the treatment period. Efficacy assessments will include the UTISA (Urinary Tract Infection Symptoms Assessment Questionnaire) together with a global assessment by the investigator. Safety assessments will include monitoring of adverse events and laboratory tests carried out at each of the three study visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, age ≥18
* Clinical diagnosis of recurrent cystitis (≥ 2 episodes in the past 6 months)
* Female subject of reproductive age not pregnant, agrees to use birth control during study period
* Subject has read, understood, signed and dated informed consent document

Exclusion Criteria:

* History of nephritis or kidney stones
* History of hepatic or gastrointestinal disease
* Diabetes
* Glaucoma
* Female subjects: pregnancy or breastfeeding
* History of anatomical alterations contributing to recurring cystitis on imaging exams
* Hypersensitivity to any component of study drug

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2018-03-31 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Urination regularity | Following three days of treatment with urinary antiseptics
  Percentage of subjects presenting improvement in cystitis symptoms in the "Urination Regularity" domain of the UTISA at Visit 2.

SECONDARY OUTCOMES:
Total UTISA score | From pretreatment to final visit, total of 6 days of treatment
  Evolution of total UTISA score at end of study compared to pretreatment in each treatment group
UTISA question # 9 | At Visit 2, after 3 days of treatment
  Percentage of subjects with improvement in UTISA question 9 at Visit 2 in each treatment group
Adverse events | From pretreatment to final visit, total of 6 days of treatment
  Incidence of study drug-related adverse events in each treatment group
Problems with Urination at Visit 2 | After 3 days of treatment
  Evolution of UTISA domain "Problems with Urination" in each treatment Group
Problems with Urination at Visit 3 | After 6 days of treatment
  Evolution of UTISA domain "Problems with Urination" in each treatment Group
Pain Associated with UTI at Visit 2 | After 3 days of treatment
  Evolution of UTISA domain "Pain Associated with UTI" in each treatment Group
Pain Associated with UTI at Visit 3 | After 6 days of treatment
  Evolution of UTISA domain "Pain Associated with UTI" in each treatment Group
Blood in Urine at Visit 2 | After 3 days of treatment
  Evolution of UTISA domain "Blood in Urine" in each treatment Group
Blood in Urine at Visit 3 | After 6 days of treatment
  Evolution of UTISA domain "Blood in Urine" in each treatment Group

CONTACTS AND LOCATIONS:
Overall Officials: carlos p nunes, MD, Principal Investigator — Fundação Educacional Serra dos Órgãos
Locations (1):
- Centro Universitário Serra dos Órgãos - UNIFESO, Teresópolis, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No